CLINICAL TRIAL: NCT02031627
Title: Physiologic Response to Varying Lymphoedema Compression Programs With the Flexitouch System
Brief Title: Treatment Response to Different Lymphoedema Compression Programs Using a Pneumatic Compression Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tactile Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4010 FlexDose
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Results first posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Lower Extremity Lymphoedema; Leg Lymphoedema
Keywords: lymphedema; lymphoedema; leg lymphoedema; lower extremity lymphoedema; pneumatic compression device
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- pneumatic compression - 1 hour per day (Experimental): Pneumatic compression device - 12 consecutive days undergoing a 1 hour treatment regimen.
  Interventions: Device: pneumatic compression - 1 hour per day
- pneumatic compression - 2 hours per day (Experimental): Pneumatic compression device - 5 consecutive days undergoing 1 hour treatment in the am and 1 hour of treatment in the pm.
  Interventions: Device: pneumatic compression - 2 hours per day
- pneumatic compression - 4 hours per day (Experimental): Pneumatic compression device - 5 consecutive days undergoing treatment twice per day consisting of 2 consecutive 1 hour treatments in the am and the pm (4 hours total)
  Interventions: Device: pneumatic compression - 4 hours per day

INTERVENTIONS:
Device: pneumatic compression - 1 hour per day — Pneumatic compression treatment once per day (1 hour)
  Other Names: Flexitouch pump; Flexitouch device
  Arms: pneumatic compression - 1 hour per day
Device: pneumatic compression - 2 hours per day — pneumatic compression treatment twice per day in the AM & PM (2 hours)
  Other Names: Flexitouch pump; Flexitouch device
  Arms: pneumatic compression - 2 hours per day
Device: pneumatic compression - 4 hours per day — pneumatic compression treatment twice per day consisting of 2 consecutive 1 hour treatments in the AM & PM (4 hours)
  Other Names: Flexitouch pump; Flexitouch device
  Arms: pneumatic compression - 4 hours per day

SUMMARY:
Proof of principle study in order to determine if there is a difference in treatment effect across the 3 study groups when treating lower extremity lymphoedema using a pneumatic compression device.

DETAILED DESCRIPTION:
This is a single center, 3 arm, prospective, randomized, clinical trial to assess the difference between 3 treatment options for achieving a measurable physiologic effect on lower extremity lymphedema with pneumatic compression device. Each intervention arm will include 10 completed subjects for a total of 30 completed subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be ≥ 18 years old
* Subjects must have a diagnosis of primary or secondary Stage 2 unilateral or bilateral lower extremity lymphoedema
* Must currently be using adequate compression garment(s) as determined by the clinician: (Garments must be at least 20mmHg and no more than 3 months old and must be worn upon rising and removed at bedtime)
* Subjects must have clinically relevant excess limb swelling as determined by clinician "pitting test"
* Must be able to attend all required in-clinic treatment visits

Exclusion Criteria:

* Diagnosis of active or recurrent cancer, or less than 3 months at the time of initial evaluation from the completion of chemotherapy, radiation therapy, or primary surgery for the treatment of cancer
* Active infection or inflammation
* Active thrombophlebitis (within the last 2 months)
* History of pulmonary embolism (within the last 2 months)
* Documented history of deep chronic venous insufficiency or deep venous obstruction with a reflux duration of > 2 second in the deep system or any history of deep vein thrombosis (DVT)
* History of pulmonary edema
* History of congestive heart failure
* History of chronic kidney disease with a glomerular filtration rate (GFR) of less than 30 mls per minute
* Poorly controlled asthma
* Symptomatic or severe peripheral artery disease (defined by current lifestyle-limiting claudication or critical limb ischemia)
* Presence of an open wound or ulcer of any etiology
* Diagnosis of lipoedema and lipolymphoedema
* Currently using an in-home pneumatic compression device
* Metal implant(s) that would interfere with bioimpedance equipment
* Pacemaker or other implanted electronic device(s)
* Unable or unwilling to remove bandaging from treatment regimen while participating in the study
* Pregnant
* Any condition where increased venous and lymphatic return is undesirable
* Unable or unwilling to participate in all aspects of the study protocol and/or unable to provide informed consent
* Currently participating in another clinical trial
* Currently using diuretics
* BMI > 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-11-11 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vaughan Keeley, PhD, FRCP, Principal Investigator — Royal Derby Hospital
Locations (1):
- Royal Derby Hospital, Derby, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: 12 consecutive days undergoing a 1-hour pneumatic compression treatment once per day (1 hour total daily)
- Group B: 5 consecutive days undergoing a 1-hour pneumatic compression treatment in the AM and 1 hour of treatment in the PM (2 hours total daily)
- Group C: 5 consecutive days undergoing 2 consecutive 1-hour pneumatic compression treatments in the AM and again in the PM (4 hours total daily)
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 7 | 7 | 7
Completed | 7 | 7 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 7 | 7 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (6.7) | 58.1 (11.1) | 50.4 (18.3) | 58.0 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 6 | 18
  Male | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 7 | 7 | 6 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 7 | 7 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Limb Volume (ml)
Description: Limb volume changes measured via perometry reported in change of ml of fluid. A negative value is associated with the clinically-desirable decrease in fluid.
Time Frame: Change baseline to final day (day 12 for Group A and day 5 for Groups B and C)
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 7 | 7
ml | -197 (78) | -60 (126) | 45 (381)

2. Primary Outcome: Limb Volume (% Change)
Description: Limb volume changes measured via perometry reported in percent reduction. A negative value is associated with the clinically-desirable decrease in fluid.
Time Frame: Change baseline to final day (day 12 for Group A and day 5 for Groups B and C)
Measure: Mean (Standard Deviation); unit: % reduction
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 7 | 7
% reduction | -2.6 (1.1) | -0.7 (1.3) | 0.6 (4.5)

3. Primary Outcome: Change in Skin Tone
Description: Change in skin tone (fibrosis) measured via tonometry. The tonometer is a mechanical device that gives an indication of the resistance of tissue to compression. It is used in lymphedema to give an estimate of the extent of pitting and fibrotic induration. Tonometry measures were collected at 5 anatomical locations. A negative value is associated with a clinically desirable decrease in tone.
Time Frame: Change baseline to final day (day 12 for Group A and day 5 for Groups B and C)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 7 | 7
mm
  Dorsum of Central Foot | 0.1 (0.7) | 0.5 (2.0) | 0.2 (1.1)
  Posterior to Medial Malleolus | -0.3 (1.6) | -0.7 (3.6) | -1.2 (3.3)
  7 cm From Bottom of Patella (along midline) | -0.6 (1.5) | 0.2 (2.0) | 0.8 (1.1)
  7 cm From Top of Patella (along midline) | -0.3 (1.2) | -0.7 (3.6) | -0.1 (1.1)
  7 cm Below Inguinal Crease (along midline) | -0.2 (5.0) | -0.9 (3) | -0.8 (2.1)
  Abdominal Wall (7 cm below umbilicus) | 0.3 (0.5) | -0.7 (2.4) | 0.3 (0.5)

4. Primary Outcome: Patient Reported Outcomes - MYMOP
Description: Changes in patient-determined symptoms* and change in affect the symptoms had on the subject. Measured via MYMOP (Measure Yourself Medical Outcome Profile) questionnaire. A low score indicates a good outcome. Scores range from 0 (as good as can be) to 6 (as bad as can be).
  *Recorded symptoms were: Gr A, 1st symptom: none, abdominal pain and discomfort, swelling, physical, and worrying about granddaughters Gr B, 1st symptom: arthritis, hayfever, look of fat foot, right hand area of neck and shoulder, stairs, and swelling Gr C, 1st symptom: none, energy during dancing and gardening, frustration of not going out on own, swelling, mild longstanding depression, and MPT joint at base of small toe Gr A, 2nd symptom: fatigue, heaviness of leg, mental, and pain under knee Gr B, 2nd symptom: narrowed choice of footwear, shower in bath, and swollen left foot Gr C, 2nd symptom: being tired and aching all over, and shoes and clothing
Time Frame: Change baseline to final day (day 12 for Group A and day 5 for Groups B and C)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 7 | 7
score on a scale
  First Symptom (see Outcome Measure Description) | -1.8 (1.9) | -0.7 (0.8) | -0.3 (1.3)
  Second Symptom (see Outcome Measure Description) | -1.3 (1.2) | 0 (0) | -1.5 (0.7)
  Activity | -1.4 (0.9) | -1.0 (1.7) | -0.5 (0.7)
  Well-Being | -0.8 (1.3) | -0.3 (1.8) | 0 (0)

5. Secondary Outcome: Cellular Fluid Changes (Ohms)
Description: Changes in extra cellular fluid (ECF) on treated leg measured by bioimpedance. A negative number is indicative of a clinically desirable reduction in ECF.
Time Frame: Change after initial treatment on day 1 and change baseline to end of day 5 for all groups
Measure: Mean (Standard Deviation); unit: ohms
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 7 | 7
ohms
  ECF change following initial treatment (ohms) | -5.8 (17.4) | -12.1 (19.0) | -3.8 (15.1)
  ECF change from baseline to end of day 5 (ohms) | -12.3 (22) | -4.6 (27.2) | 2.1 (24.5)

6. Secondary Outcome: Cellular Fluid Changes (% Change)
Description: as for outcome 5
Time Frame: Change after initial treatment on day 1 and change baseline to end of day 5 for all groups
Measure: Mean (Standard Deviation); unit: percent fluid change
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 7 | 7
percent fluid change
  ECF change following initial treatment (percent) | -2.5 (6.9) | -4.5 (6.4) | -1.2 (6.6)
  ECF change from baseline to end of day 5 (percent) | -4.9 (8.0) | -2.0 (10.5) | 1.1 (11.9)

7. Secondary Outcome: Incidence of Complications
Description: Number of complications experienced. Incidence based on clinician assessment.
Time Frame: Change baseline to final day (day 12 for Group A and day 5 for Groups B and C)
Measure: Number; unit: Complications
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 7 | 7
Complications | 0 | 0 | 0

8. Secondary Outcome: Activity Level
Description: Change in number of steps as accumulated each day monitored through use of a pedometer. A positive number indicates an increase in step count (activity) while a negative number indicates a decrease in step count.
Time Frame: Day 1 compared to final treatment day (day 12 for Group A and day 5 for Groups B and C)
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 7 | 7
steps | 28 (281) | -1284 (2144) | 1240 (1916)

9. Other Pre Specified Outcome: Change in Skin Thickness
Description: Change in skin thickness measured by ultrasound. Ultrasound measures were collected at 5 anatomical locations. A negative value is associated with a clinically desirable reduction in skin thickness (a surrogate measure of oedema).
Time Frame: Change baseline to final day (day 12 for Group A and day 5 for Groups B and C)
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 7 | 7
cm
  Dorsum of Central Foot | -0.09 (0.13) | 0.02 (0.11) | -0.02 (0.04)
  Posterior to Medial Malleolus | 0.12 (0.13) | -0.06 (0.16) | 0.04 (0.12)
  7 cm From Bottom of Patella (along midline) | -0.02 (0.08) | 0.00 (0.07) | -0.03 (0.02)
  7 cm From Top of Patella (along midline) | -0.01 (0.02) | -0.01 (0.04) | 0.00 (0.05)
  7 cm Below Inguinal Crease (along midline) | -0.01 (0.05) | -0.01 (0.05) | 0.00 (0.03)
  Abdominal Wall (7 cm below umbilicus) | -0.01 (0.04) | 0.00 (0.04) | -0.02 (0.04)

10. Other Pre Specified Outcome: Change in Local Tissue Water (LTW)
Description: Change in local tissue water (LTW) within the skin measured by MoistureMeterD (MMD). MMD measures were collected at 5 anatomical locations using 2 probes: medium (M25) and large (L50). A negative value is associated with a clinically desirable decrease in LTW (a surrogate measure of oedema).
Time Frame: Change baseline to final day (day 12 for Group A and day 5 for Groups B and C)
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 7 | 7
cm
  M25 Probe: Dorsum of Central Foot | 1.9 (5.8) | -1.1 (5.4) | 2.9 (10.8)
  L50 Probe: Dorsum of Central Foot | 6.4 (10.6) | -6.3 (9.6) | -0.9 (10.4)
  M25 Probe: Posterior to Medial Malleolus | 2.5 (6.0) | 3.2 (4.5) | 4.7 (6.0)
  L50 Probe: Posterior to Medial Malleolus | -2.3 (5.4) | 3.4 (9.0) | 2.5 (6.3)
  M25 Probe: 7 cm From Bottom of Patella (along midline) | 2.3 (5.6) | 0.6 (5.5) | 2.0 (5.8)
  L50 Probe: 7 cm From Bottom of Patella (along midline) | 3.4 (6.9) | -0.3 (3.5) | 0.1 (6.4)
  M25 Probe: 7 cm From Top of Patella (along midline) | 1.3 (1.6) | 2.4 (1.4) | 3.1 (4.4)
  L50 Probe: 7 cm From Top of Patella (along midline) | -0.8 (1.6) | -0.2 (1.8) | 3.2 (4.6)
  M25 Probe: 7 cm Below Inguinal Crease (along midline) | 1.3 (3.7) | 2.0 (2.1) | 0.9 (3.0)
  L50 Probe: 7 cm Below Inguinal Crease (along midline) | -1.2 (1.5) | 1.3 (0.7) | 0.6 (1.9)
  M25 Probe: Abdominal Wall (7 cm below umbilicus) | 0.9 (3.6) | 0.9 (1.8) | 1.3 (5.3)
  L50 Probe: Abdominal Wall (7 cm below umbilicus) | -0.1 (1.4) | -1.1 (2.7) | 0.2 (1.6)

11. Post Hoc Outcome: Patient Reported Outcomes - LYMQOL
Description: Self-reported changes in symptoms in 4 domains: function, appearance, symptoms, and emotion as well as general quality of life (QOL). Measured via LYMQOL (Lymphedema Quality of Life) questionnaire. A decrease in the the domain scores and increase in general QOL indicate a good outcome. Scores range from 1 to 4.
Time Frame: Change baseline to final day (day 12 for Group A and day 5 for Groups B and C)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 7 | 7
score on a scale
  Function | -2.2 (2.4) | -0.8 (2.9) | 0.1 (3.4)
  Appearance | -4.2 (6.1) | -0.6 (4.0) | -0.2 (4.4)
  Symptoms | -3.0 (4.0) | -1.6 (2.9) | -2.2 (4.5)
  Emotion | -1.4 (3.1) | -1.0 (5.2) | 0.5 (1.6)
  Overall Quality of Life (QOL) | -0.7 (0.5) | -0.7 (1.5) | 0.3 (0.8)

ADVERSE EVENTS:
Time Frame: 12 days after baseline for Group A, 5 days after baseline for Groups B and C
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-13): https://cdn.clinicaltrials.gov/large-docs/27/NCT02031627/Prot_SAP_000.pdf